CLINICAL TRIAL: NCT03781063
Title: An Open-Label, Randomized, Multicenter Study Evaluating the Activity of Lasofoxifene Relative to Fulvestrant for the Treatment of Pre- and Postmenopausal Women With Locally Advanced or Metastatic ER+/HER2- Breast Cancer With an ESR1 Mutation
Brief Title: Evaluation of Lasofoxifene Versus Fulvestrant in Advanced or Metastatic ER+/HER2- Breast Cancer With an ESR1 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sermonix Pharmaceuticals Inc. (Industry)
Collaborators: Linical Accelovance Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMX 18001
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: Locally Advanced Breast Cancer; Metastatic Breast Cancer; Lasofoxifene; Fulvestrant; ER+/HER2; ESR1 mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — Lasofoxifene; Fulvestrant

STUDY DESIGN:
Intervention Model Description: open label, randomized, parallel-group, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lasofoxifene (Experimental): 5 mg/d of oral lasofoxifene
  Interventions: Drug: Lasofoxifene
- Fulvestrant (Active Comparator): 500 mg fulvestrant intramuscular (IM)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Lasofoxifene — Estrogen receptor antagonist antineoplastic agent
  Arms: Lasofoxifene
Drug: Fulvestrant — Estrogen receptor antagonist antineoplastic agent
  Arms: Fulvestrant

SUMMARY:
This is an open label, randomized, multicenter study evaluating the activity of lasofoxifene relative to fulvestrant for the treatment of pre- and postmenopausal women with locally advanced or metastatic ER+/HER2- breast cancer with an acquired ESR1 mutation and who have disease progression on an aromatase inhibitor (AI) in combination with a cyclin dependent kinase (CDK) 4/6 inhibitor.

The primary objective is to evaluate the progression free survival (PFS) of 5 mg lasofoxifene relative to fulvestrant for the treatment of pre- and postmenopausal women with locally advanced or metastatic estrogen receptor positive (ER+)/human epidermal growth factor 2 negative (HER2-) breast cancer with an estrogen receptor 1 (ESR1) mutation.

The secondary objectives are to evaluate:

1. Clinical benefit rate (CBR) and Objective Response Rate (ORR)
2. Duration of response
3. Time to response
4. Overall Survival (OS)
5. Pharmacokinetics of lasofoxifene
6. Quality of life (QoL): Quality of Life (QoL): vaginal assessment scale (VAS) and vulvar assessment scale (VuAS) questionnaires
7. Safety of lasofoxifene
8. Response to various ESR1 mutation (Y537S, Y537C, D538G, E380Q, S463P, V534E, P535H, L536H, L536P, L536R, L536Q, or Y537N).

DETAILED DESCRIPTION:
Lasofoxifene is a potent SERM that has demonstrated in non-clinical models to prevent and treat breast cancer. In a large clinical osteoporosis trial, lasofoxifene reduced the incidence of ER+ breast cancer, which most likely represents a beneficial effect on clinically undetectable breast cancer. The clinical and non-clinical results are not unexpected based on the results seen with tamoxifen and fulvestrant as the mechanisms of action are similar. Moreover, the safety profile of lasofoxifene is well established in postmenopausal women and therefore a clinical trial investigating lasofoxifene for the treatment of breast cancer is scientifically justifiable.

Subjects with ESR1 mutations have endocrine resistance and shorter time to progression when treated with currently approved endocrine therapy. There is an unmet medical need for endocrine agents that can provide greater efficacy in this population. Non-clinical in vitro and in vivo studies with lasofoxifene have demonstrated efficacy. If this benefit translates to subjects with ESR1 mutated breast cancer cells, an important treatment option beyond fulvestrant will be available. The population being recruited in this trial are subjects with advanced breast cancer who have been treated with an AI in combination with a cyclin-dependent kinase (CDK) 4/6 inhibitor and who have an ESR1 mutation. The efficacy of endocrine agents in this population has never been prospectively studied. For this reason, this study will evaluate lasofoxifene in a randomized Phase 2 trial against a comparator to better evaluate the magnitude of the effect as well as to provide data to estimate the Phase 3 sample size.

In both non-clinical and clinical studies, fulvestrant has shown activity in ESR1 mutated breast cancer cells and will be used as the comparator in this Phase 2 study to better determine the relative clinical efficacy of lasofoxifene. The FDA approved fulvestrant dose will be used.

A major limiting factor in the administration of fulvestrant is its poor solubility requiring IM injection. The volume of administration limits the dose that can be administered. Initial clinical trials administered 250 mg of fulvestrant in 5 cc of castor oil as a single injection once monthly. Because the IM injections were well tolerated, loading and higher doses were investigated. This was found to have acceptable tolerability and resulted in greater efficacy. Limited by the volume of administration higher doses of fulvestrant cannot be investigated further.

Once the subject has consented to participate in the study, screening tests will be performed within 30 days of enrollment.

All subjects meeting the eligibility criteria will be first stratified into those with visceral metastasis and those without visceral metastasis. Each of these stratified groups will then be further stratified into those with the Y537S ESR1 mutation and those without this particular mutation. Each of the stratified groups will then be randomized 1:1 to receive either 5 mg/d of oral lasofoxifene or fulvestrant 500 mg intramuscular (IM) on Days 1, 15, and 29, then every 4 weeks thereafter. Treatment will continue until radiographic or clinical evidence of disease progression. Enrolled subjects will be seen every 2 weeks for the first month of treatment and then monthly until progression. Efficacy assessments will be done every 8 weeks.

For subjects randomized to lasofoxifene, blood samples will be drawn to assess the population PK. Serum samples will be collected at each visit starting at Visit 0 (Day 1) through Final/ET visit to measure serum lasofoxifene concentration at time points outlined below. Serum samples for PK analysis will be collected before the time that the next lasofoxifene dose is ingested. The actual time and date of dosing on the previous day as well as dosing on the visit day, and the PK blood sampling time/date must be recorded for all subjects. Pharmacokinetic samples are to be collected before clinical lab blood sampling.

A maximum of 100 subjects will be randomized and it is expected that all subjects enrolled in the study will be treated until documented disease progression. It is estimated that full recruitment into the study will occur within 12 to 18 months with another 12 months of follow up before the primary outcome measure is analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or postmenopausal.

   Postmenopausal women are defined as:
   1. ≥60 years of age with no vaginal bleeding over the prior year, or
   2. <60 years with "premature menopause" or "premature ovarian failure" manifest itself with secondary amenorrhea for at least 1 year and follicle stimulating hormone (FSH) and estradiol levels in the postmenopausal range according to institutional standards, or
   3. surgical menopause with bilateral oophorectomy. Note: premenopausal women who meet all of the other entry criteria must be maintained on ovarian suppression (such as Lupron) during the study and subjects counseled to use appropriate contraception to prevent pregnancy.
2. If possible, a biopsy of metastatic breast cancer tissue will be obtained to provide histological or cytological confirmation of ER+ and HER2- disease as assessed by a local laboratory, according to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines, using slides, paraffin blocks, or paraffin samples. If a biopsy is not possible, the ER and HER2 status from the tissue obtained at the time of the original diagnosis must confirm that the subject's cancer is ER+ and HER2-.
3. Locally advanced or metastatic breast cancer with radiological or clinical evidence of progression on an AI in combination with a CDK 4/6 inhibitor for advanced breast cancer with demonstrated prior sensitivity to endocrine therapy (recurrence or progression after at least 12 months of treatment in the metastatic setting).
4. Locally advanced or metastatic breast cancer with either measurable (according to RECIST 1.1) or non-measurable lesions.
5. At least one or more of the following point ESR1 mutations as assessed in cell-free circulating tumor DNA (ctDNA) obtained from a blood (plasma) or tissue sample: Y537S, Y537C, D538G, E380Q, S463P, V534E, P535H, L536H, L536P, L536R, L536Q, or Y537N. The ctDNA sample collection must be obtained within 30 days prior to randomization to determine eligibility and baseline. Note: a prior genomic test confirming that the subject has an ESR1 mutation can be used to determine eligibility; however, an ESR1 sample must also be collected within 30 days of randomization.
6. Subjects who have not received cytotoxic chemotherapy or those who have received one cytotoxic chemotherapy regimen in the neo-adjuvant or adjuvant setting prior to entry into the trial and/or no more than one chemotherapy regimen for metastatic breast cancer. Subjects must be free of all chemotherapy acute toxicity excluding alopecia and Grade II peripheral neuropathy before study entry.
7. ECOG performance score of 0 or 1.
8. Adequate organ function as shown by:

   1. absolute neutrophil count (ANC) >/=1,500 cells/mm3
   2. platelet count ≤100,000 cells/mm3
   3. hemoglobin >/=9.0 g/dl
   4. ALT and AST levels ≤2.5 upper limit of normal (ULN) or ≤5 in the presence of visceral metastasis
   5. total serum bilirubin ≤1.5 X ULN (≤ 3 X ULN for subjects known to have Gilbert Syndrome)
   6. alkaline phosphatase level ≤ 2.5 X ULN
   7. creatinine clearance of 40 ml/min or greater as calculated by the Cockcroft-Gault formula
   8. International normalized ratio (INR), activated partial thromboplastin (aPTT), or partial thromboplastin time (PTT) <2.0 X ULN.
9. Able to swallow tablets.
10. Able to understand and voluntarily sign a written informed consent before any screening procedures.

Exclusion Criteria:

1. Prior use of everolimus or other mammalian target of rapamycin (mTOR) inhibitor or phosphoinositide 3-kinase inhibitor (PI3K) inhibitors is excluded unless discontinued to reasons other than disease progression.
2. Presence of brain metastasis.
3. Lymphangitic carcinomatosis involving the lung.
4. Impending visceral crisis in need of cytotoxic chemotherapy as assessed by the investigator.
5. Radiotherapy within 30 days prior to randomization except in case of localized radiotherapy for analgesic purposes or for lytic lesions at risk of fracture, which can then be completed within 7 days prior to randomization. Subjects must have recovered from radiotherapy toxicities prior to randomization.
6. History of long QTC syndrome or a QTC of >480 ms.
7. History of a pulmonary embolus (PE) or deep vein thrombosis (DVT) within the last 6 months or any known thrombophilia. Subjects stable on anti-coagulants for maintenance are eligible as long as the DVT and/or PE occurred >6 months prior to enrollment and there is no evidence for active thrombosis. The use of low dose ASA is permitted.
8. Any significant co-morbidity that would impact the study or the subject's safety.
9. History of a positive human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) at Screening. Subjects cured of hepatitis C (no viral load) are eligible.
10. History of malignancy within the past 5 years (excluding breast cancer), except basal cell or squamous cell carcinoma of the skin curatively treated by surgery, or early stage cervical cancer.
11. History of vaginal bleeding over the last year unless it is documented that the bleeding was due to non-uterine causes (e.g. vaginal atrophy).
12. Uncontrolled hypertension defined as sitting systolic pressure >160 mm Hg or diastolic pressure >100 mm Hg at Screening.
13. History of non-compliance to medical regimens.
14. Unwilling or unable to comply with the protocol.
15. Current participation in any clinical research trial involving an investigational drug or device within the last 30 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre- and Postmenopausal women
Enrollment: 100 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, an average of 1 year
  PFS is defined as the interval from the date of randomization to the earlier date of first documented radiographic progression or death due to any cause

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | through study completion, an average of 1 year
  CBR is defined as the percentage of all subjects with a complete or partial response; or stable disease for >/=24 weeks.
Objective Response Rate (ORR) | through study completion, an average of 1 year
  ORR is defined as the percentage of subjects with either a complete response (CR) or a partial response (PR) as assessed by the RECIST 1.1 criteria.
Overall Survival (OS) | through study completion, an average of 1 year
  OS is defined as time from randomization to death due to any cause.
Incidence of Adverse Events (AEs) and Serious AEs | through study completion, an average of 1 year
  The type, severity (graded by Common Terminology Criteria for Adverse Events [CTCAE version 5.0]), course, duration, seriousness, and relationship to study treatment will be assess at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul V. Plourde, MD, Study Director — Sermonix Pharmaceuticals
Locations (51):
- United States (42):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Yuma Regional Medical Center (JIT), Yuma, Arizona
  - City of Hope Comprehensive Cancer, Duarte, California
  - Compassionate Care Research Group, Fountain Valley, California
  - UCSF Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Ocala Oncology Center (JIT), Oscala, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - The Bond Clinic Cancer & Research Center., Winter Haven, Florida
  - Emory University, Atlanta, Georgia
  - Hawaii Cancer Care (JIT), Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Illinois Cancer Care (JIT), Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Beacon Health (JIT), South Bend, Indiana
  - University of Louisville / James Graham Brown Cancer Center, Louisville, Kentucky
  - FMH James M Stockman Cancer Institute (JIT), Frederick, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - HCA Midwest Health, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada (JIT), Las Vegas, Nevada
  - New Jersey Cancer Care and Blood Disorders (JIT), Belleville, New Jersey
  - Summit Medical Group (JIT), Florham Park, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - The Ohio State University - Comprehensive Cancer Center, Columbus, Ohio
  - Ohio Health (JIT), Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sanford Cancer Center (JIT), Sioux Falls, South Dakota
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology/SCRI, Nashville, Tennessee
  - Mary Crowley Cancer Research (JIT), Dallas, Texas
  - Oncology Consultants (JIT), Houston, Texas
  - Utah Cancer Specialists (JIT), Salt Lake City, Utah
  - Peninsula Cancer Institute, Newport News, Virginia
- Canada (5):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - CIUSSS de Saguenay-Lac-Saint Jean, Chicoutimi, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Israel (4):
  - Soroka University Medical Center, Beersheba, Israel
  - Hadassah Ein Kerem Medical Center, Jerusalem, Israel
  - Rabin Medical Center, Petah Tikva, Israel
  - Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Goetz MP, Bagegni NA, Batist G, Brufsky A, Cristofanilli MA, Damodaran S, Daniel BR, Fleming GF, Gradishar WJ, Graff SL, Grosse Perdekamp MT, Hamilton E, Lavasani S, Moreno-Aspitia A, O'Connor T, Pluard TJ, Rugo HS, Sammons SL, Schwartzberg LS, Stover DG, Vidal GA, Wang G, Warner E, Yerushalmi R, Plourde PV, Portman DJ, Gal-Yam EN. Lasofoxifene versus fulvestrant for ER+/HER2- metastatic breast cancer with an ESR1 mutation: results from the randomized, phase II ELAINE 1 trial. Ann Oncol. 2023 Dec;34(12):1141-1151. doi: 10.1016/j.annonc.2023.09.3104. PMID 38072514